CLINICAL TRIAL: NCT00274703
Title: A Randomised, Double-Blind, Placebo-Controlled, Single-Centre Study to Provide a Preliminary Evaluation of Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Intravenous Anti-human Interleukin-5 (Mepolizumab, 750mg and 1500mg) in the Treatment of Eosinophilic Oesophagitis in Adults
Brief Title: An Evaluation Of Mepolizumab In Therapy Of Eosinophilic Oesophagitis In Adult Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MEE103226
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Oesophagitis, Eosinophilic
Keywords: anti IL-5; oesophagitis; eosinophils; mepolizumab; adults
MeSH Terms: conditions — Esophagitis | interventions — mepolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: mepolizumab

SUMMARY:
Eosinophils play a key role in the pathogenesis of eosinophilic oesophagitis. Therapies that suppress eosinophil recruitment and activation may give a benefit. Mepolizumab is a humanised monoclonal antibody against interleukin-5 (IL-5). This study will evaluate the ability of mepolizumab to decrease the recruitment and infiltration of eosinophils into the oesophagus, thereby reducing the inflammation and symptoms of EE (eosinophilic oesophagitis) in adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Document evidence/presence of Oesophagitis prior to commencing trial drug.
* a)Histological evidence of Oesophagitis: greater than 20x eosinophils per high power field (X400) on histology of esophageal mucosal biopsy
* b. at least one episode of dysphagia per week
* c.Inadequate response to routine EE treatment
* D. No other known causes of oesophagitis, or esophageal or generalized eosinophilia
* Not pregnant or nursing

Exclusion criteria:

* History of seasonal worsening of EE symptoms or requirement of Esophageal dilation.
* Churg-Strauss Syndrome
* Wegener's Granulomatosis
* Lymphoma, hematological malignancy, advanced and metastatic solid tumors
* Active H. pylori infection.
* Any previous treatment with anti-hIL-5, anti-IgE monoclonal antibody or other biological agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-12; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
1. Reduction of eosinophils in the oesophagus 2. Safety and tolerability of mepolizumab

SECONDARY OUTCOMES:
1. Effect of treatment on symptoms, Eosinophil levels, and on inflammation biomarkers in oesophagus tissue and blood.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Olten, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Conus S, Straumann A, Bettler E, Simon HU. Mepolizumab does not alter levels of eosinophils, T cells, and mast cells in the duodenal mucosa in eosinophilic esophagitis. J Allergy Clin Immunol. 2010 Jul;126(1):175-7. doi: 10.1016/j.jaci.2010.04.029. Epub 2010 Jun 12. No abstract available. PMID 20542323
- [Derived] Straumann A, Conus S, Grzonka P, Kita H, Kephart G, Bussmann C, Beglinger C, Smith DA, Patel J, Byrne M, Simon HU. Anti-interleukin-5 antibody treatment (mepolizumab) in active eosinophilic oesophagitis: a randomised, placebo-controlled, double-blind trial. Gut. 2010 Jan;59(1):21-30. doi: 10.1136/gut.2009.178558. PMID 19828470
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: MEE103226 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: MEE103226 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: MEE103226 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: MEE103226 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: MEE103226 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register